CLINICAL TRIAL: NCT07163611
Title: Obinutuzumab Induced Decreases of PLA2Rab in MN: a Pilot Study
Brief Title: Obinutuzumab Induced Decreases of PLA2R Antibodies in Membranous Nephropathy: a Pilot Study
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-521139-35-01; 2025-521139-35-01 (EU CTIS Number)
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: Membranous Nephropathy - PLA2R Induced
Keywords: PLA2R antibody kinetics; membranous nephropathy; obinutuzumab
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with obinutuzumab. (Experimental)
  Interventions: Drug: Obinutuzumab administration

INTERVENTIONS:
Drug: Obinutuzumab administration — All participants will receive obinutuzumab 1000 mg on day 1 and 15, with two additional infusions after 6 months if the anti-PLA2R antibody IFT assay is still positive with proteinuria > 2 gram/24 hours and stable kidney function.

SUMMARY:
Objective: To assess the disappearance rate (half-life) of anti-PLA2R antibodies in high-risk primary membranous nephropathy (pMN) patients treated with obinutuzumab (OBI), and to evaluate immunological and clinical remission, adverse events, and quality of life.

Design: Open-label, single-center, prospective pilot intervention study conducted at Radboud University Medical Center.

Population: 20 adult patients with high-risk PMN, defined by proteinuria ≥3.5 g/24h despite 6 months of supportive treatment with ACE inhibitors or ARBs.

Intervention: OBI 1000 mg on days 1 and 15, with two additional infusions after 6 months if anti-PLA2R antibody levels remain positive and proteinuria exceeds 2 g/24h.

Follow-up: Patients were monitored at baseline, and at weeks 1, 2, 4, 8, 12, 24, 37, and 52.

DETAILED DESCRIPTION:
Rationale:

Primary membranous nephropathy (PMN) is a leading cause of nephrotic syndrome in adults and is characterized by subepithelial immune complex deposits in the glomerular basement membrane. The disease is associated with circulating auto-antibodies targeting the M-type phospholipase A2 receptor (PLA2R), present in 70-80% of patients.

Despite advances in understanding its pathogenesis, the optimal treatment of PMN remains suboptimal; as the response to immunosuppressive therapy is often limited and slow. When considering treatment in PMN, the overall response rate is important, but in high-risk PMN patients the rapidity of response is even more important. As so, ideally we should be able to identify non-responders and slow-responders before or within a few months after start of therapy. A regimen consisting of rituximab (RTX), cyclophosphamide (CP) and steroids (triple therapy) has proven that a rapid immunological and clinical remission in PMN patients is possible. Obinutuzumab (OBI), a next-generation fully humanized anti-CD20 monoclonal antibody, offers enhanced B cell depletion through greater antibody-dependent cytotoxicity and reduced complement activation when compared to RTX. Retrospective studies suggests that OBI demonstrates superior efficacy in the treatment of treatment-refractory PMN patients compared to RTX, while maintaining a similar safety profile. It has been proven effective in the treatment of proliferative lupus nephritis compared to standard-of-care. These studies not only suggested better overall response, but the data also indicated a more rapid onset of remission.

Objective:

The primary objective of this pilot study is to calculate disappearance rate (half-life) of anti-PLA2R antibodies in PMN patients treated with OBI. We hypothesize that OBI monotherapy might be able to induce a rapid immunological response comparable to triple therapy in high-risk PLA2Rab-associated PMN patients. Secondary outcome measures are immunological remission, complete or partial clinical remission, adverse events and quality of life.

Main trial endpoint:

The main trial endpoint is the disappearance rate (half-life) of anti-PLA2R antibodies in PMN patients after treatment with OBI.

Secondary trial endpoints:

Immunological remission defined as IFT negative. Efficacy on clinical disease activity, defined as either CR or PR at 12 months. Adverse events. Quality of life during OBI treatment.

Trial design:

This is an open-label single-center, prospective, pilot intervention study in the Radboud UMC hospital. Patients at our outpatient clinic with high-risk PMN, defined by proteinuria ≥ 3.5 g/24h despite supportive treatment for at least 6 months with maximally tolerated and stable dose of ACE-i or ARB without life-threatening nephrotic syndrome and/or > 20% increase in serum creatinine not otherwise explained, that are eligible for inclusion will be asked to participate in the study. A total of 20 incident and prevalent PMN patients will be included. After informed consent participants will receive OBI 1000 mg on day 1 and 15, with two additional infusions after 6 months if the PLA2Rab IFT assay is still positive with proteinuria > 2 gram/24 hours and stable kidney function.

Patients will visit our outpatient clinic at baseline, in week 1, 2, 4, 8, 12, 24, 37 and 52. During the visits to our outpatient clinic, standard measurements will be performed, including blood pressure measurement, weight monitoring and laboratory testing, including PLA2Rab monitoring. Except for week 1, in which only PLA2Rab monitoring will be conducted. The "Kidney Disease Quality of Life-36" questionnaire will be completed at baseline and in week 12, 24, 37 and 52 prior to a visit to our outpatient clinic.

Trial population:

A total of 20 adult incident and prevalent anti-PLA2R antibody-associated high-risk PMN patients will be recruited from our renal unit.

Interventions:

All participants will receive OBI 1000 mg on day 1 and 15, with two additional infusions after 6 months if the anti-PLA2R antibody IFT assay is still positive with proteinuria > 2 gram/24 hours and stable kidney function. Anti-PLA2R antibodies will be measured at baseline and week 1, 2, 4, 8, 12, 24, 37 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of PMN, confirmed by:

  1. Kidney biopsy or
  2. Positive serum PLA2Rab test either by IFT and/or ELISA)
* Serum PLA2Rab titer > 80 RU/ml
* Proteinuria ≥ 3.5 g/24h despite supportive treatment for at least 6 months with a maximally tolerated and stable dose of ACE-i or ARB.
* Serum albumin < 30 g/l measured by BCP assay.
* eGFR ≥ 30 ml/min/1.73m2.
* Treatment with immunosuppression is warranted, as determined by the treating physician.

Exclusion Criteria:

* Secondary MN (e.g., hepatitis B or C infection, human immunodeficiency virus infection, active infection, systemic lupus erythematosus, sarcoidosis, IgG4-related, drug-induced, malignancy).
* RTX within 12 months prior to inclusion.
* CNI within 2 months prior to inclusion.
* Treatment with other immunosuppressive drugs within 6 months prior to inclusion.
* Proteinuria must not have decreased by > 50% over 6 months whilst taking ACEi/ARB.
* Life-threatening nephrotic syndrome resistant to treatment.
* > 20% increase in serum creatinine not otherwise explained during antiproteinuric supportive treatment.
* Pregnancy or breastfeeding. Women of childbearing age and male patients with female partners of childbearing potential not willing to use contraception throughout the study and for at least 6 months after the last dose of obinutuzumab.
* Suspected or known hypersensitivity, allergy, and/or immunogenic reaction history to monoclonal antibodies, corticosteroid, cyclophosphamide, any of their ingredients, and any other drugs from these same pharmacotherapeutic groups.
* Known active infection of any kind or recent major episode of infection.
* Any disorder or condition which might pose an unacceptable risk to patient's safety and well-being that might interfere with completion of the study.
* Inability to understand or comply with the requirements of the study.
* Incapable of recognizing the nature, significance, and scope of the clinical trial or giving consent even with a legal representative.
* Use of an investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Disappearance rate of PLA2R antibodies | From baseline to 52 weeks after the first obinutuzumab infusion.
  To calculate the disappearance rate (half-life) of anti-PLA2R antibodies. Serum PLA2R antibodies will be measured at baseline, 1, 2, 4, 8, 12, 24 37 and 52 weeks after obinutuzumab infusions.

SECONDARY OUTCOMES:
Immunological remission | From baseline to 52 weeks after the last obinutuzumab infusion.
  Immunological remission, defined as negative accorording to the anti-PLA2R antibody immunofluorescence test (IFT).
Clinical efficacy | From baseline to 52 weeks after the last obinutuzumab infusion.
  To assess efficacy of obinutuzumab on disease activity, defined as either complete remission (CR) or partial remission (PR).
Adverse events | From baseline to 52 weeks after the last obinutuzumab infusion.
  To assess adverse events of treatment with obinutuzumab, categorized as SAE or NSAESI.
Quality of life during treatment | From baseline to 52 weeks after the last obinutuzumab infusion.
  To determine quality of life (Kidney Disease Quality of Life-36) during obinutuzumab treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Els Van de Logt, M.D., PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Department of Nephrology, Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided